CLINICAL TRIAL: NCT04047251
Title: A Phase 1 Study of FF-10850 Topotecan Liposome Injection in Advanced Solid Tumors Including Ovarian and Cervical Carcinoma, Sarcomas, and Neuroendocrine Tumors Including Small Cell Lung Cancer and Merkel Cell Carcinoma
Brief Title: A Study of FF-10850 Topotecan Liposome Injection in Advanced Solid Tumors Including Merkel Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fujifilm Pharmaceuticals U.S.A., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FF10850US101
Record Dates: First submitted 2019-08-01; First posted 2019-08-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors; Merkel Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell

STUDY DESIGN:
Intervention Model Description: Open label, dose escalation
Masking Description: None, open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: Treatment at Dose Level 1 (Experimental): FF-10850 Topotecan Liposome Injection, Dose Level 1 administered intravenously (IV) on Days 1 and 15 of each 28-day cycle
  Interventions: Drug: FF-10850 Topotecan Liposome Injection
- Cohort 2: Treatment at Dose Level 2 (Experimental): FF-10850 Topotecan Liposome Injection, Dose Level 2 administered intravenously (IV) on Days 1 and 15 of each 28-day cycle
  Interventions: Drug: FF-10850 Topotecan Liposome Injection
- Cohort 3: Treatment at Dose Level 3 (Experimental): FF-10850 Topotecan Liposome Injection, Dose Level 3 administered intravenously (IV) on Days 1 and 15 of each 28-day cycle
  Interventions: Drug: FF-10850 Topotecan Liposome Injection
- Cohort E1: Treatment at Recommended Phase 2 Dose (RP2D) (Experimental): For patients with advanced ovarian cancer: FF-10850 Topotecan Liposome Injection, RP2D administered intravenously (IV) on Days 1 and 15 of each 28-day cycle
  Interventions: Drug: FF-10850 Topotecan Liposome Injection
- Cohort E5: Treatment at Recommended Phase 2 Dose (RP2D) (Experimental): For patients with advanced Merkel cell carcinoma: FF-10850 Topotecan Liposome Injection, RP2D administered intravenously (IV) on Days 1 and 15 of each 28-day cycle
  Interventions: Drug: FF-10850 Topotecan Liposome Injection

INTERVENTIONS:
Drug: FF-10850 Topotecan Liposome Injection — FF-10850 to be diluted and infused over 60 minutes.
  Other Names: FF-10850

SUMMARY:
To determine the safety profile, maximum tolerated dose (MTD), dose-limiting toxicities (DLTs), and recommended Phase 2 dose (RP2D) of FF-10850 (topotecan liposome injection) in patients with advanced solid tumors including Merkel Cell Carcinoma

DETAILED DESCRIPTION:
Dose-escalation Phase: Approximately 48 patients are planned for the dose-escalation phase, with at least 6 patients treated at the RP2D.

Cohort Expansion Phase: Two additional cohorts are planned. Cohort E1: advanced ovarian cancer and Cohort E5 Merkel cell carcinoma. Each cohort will be treated at the RP2D.

In each cohort, FF-10850 will be administered intravenously (IV) until progression of disease, observation of unacceptable AEs, or, after discussion between the Investigator and the Medical Monitor, changes in the patient's condition that prevent further study participation. A sufficient number of cohorts will be enrolled to identify the RP2D.

There will be 3 initial dose levels in this study. FF-10850 will be diluted and infused over 60 minutes.

Approximately 96 patients are planned for the entire trial.

It is anticipated that approximately 4 centers will participate in the dose-escalation phase, with an expansion to approximately 10 centers in the cohort expansion phase. Accrual for the dose-escalation and expansion phases is expected to be approximately 3 years, with patients followed every 3 months from the last dose of study treatment to assess survival.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following criteria to participate in the study:

1. Males and females ≥ 18 years of age
2. Dose-escalation phase: Histologically or cytologically confirmed metastatic and/or unresectable solid tumor, relapsed or refractory to standard therapy, or for which no standard therapy is available that is expected to improve survival by at least 3 months
3. At least 3 weeks beyond the last chemotherapy (or 3 half-lives, whichever is shorter), radiotherapy, major surgery, or experimental treatment, and recovered from all acute toxicities (≤ Grade 1), prior to the first dose of FF-10850
4. Adequate performance status: Eastern Cooperative Oncology Group (ECOG) ≤ 1
5. Life expectancy of ≥ 3 months
6. Adequate hematologic parameters without ongoing transfusion support:

   * Hemoglobin (Hb) ≥ 9 g/dL
   * Absolute neutrophil count (ANC) ≥ 1.0 × 109 cells/L
   * Platelets ≥ 100 × 109 cells/L
7. Creatinine ≤ 1.5 × ULN, or calculated creatinine clearance ≥ 50 mL/minute by either the Cockcroft-Gault formula or as measured by a 24-hour urine collection
8. Total bilirubin ≤ 2 × ULN unless due to Gilbert's disease; patients with Gilbert's disease who have a total bilirubin > 6 mg/dL are to be excluded
9. ALT and AST ≤ 2.5 times ULN, or < 5 × ULN for patients with liver metastases
10. QT interval corrected for rate (QT interval corrected for rate using Fridericia's Correction Formula, QTcF) ≤ 470 msec for women and ≤ 450 msec for men on the ECG obtained at Screening and confirmed pre-treatment on Cycle 1 Day 1.
11. Patient must be willing to undergo a tumor biopsy, if the patient has a biopsy-accessible tumor

Exclusion Criteria:

1. Patients who have not received standard/approved therapies expected to improve survival by at least 3 months
2. History of severe hypersensitivity reactions to topotecan
3. Serious cardiac condition within the last 6 months, such as uncontrolled arrhythmia, myocardial infarction, unstable angina or heart disease defined by the New York Heart Association (NYHA) Class III or Class IV or hereditary long QT syndrome
4. Concomitant medication(s) that may cause QTc prolongation or induce Torsades de Pointes, except for antimicrobials that are used as standard of care to prevent or treat infections and other such drugs that are considered by the Investigator to be essential for patient care
5. Active central nervous system (CNS) malignant disease in patients with a history of CNS malignancy. Patients with previously treated stable brain metastases are allowed if they have been stable off steroid therapy for at least 4 weeks.
6. Known positive for human immunodeficiency virus (HIV), hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV)
7. Active infection requiring intravenous (IV) antibiotic usage within the last week prior to study treatment
8. Any other medical intervention or other condition which, in the opinion of the Principal Investigator, could compromise adherence to study requirements or confound the interpretation of study results
9. Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Determine incidence of Treatment Emergent Adverse Events | 4 years
  Safety and tolerability assessed by adverse events (AEs) and serious adverse events (SAEs)
Identify dose-limiting toxicities (DLT) of FF-10850 | 4 years
  DLT is defined as any adverse event at least possibly related to FF-10850, and meeting specified DLT criteria
Determine maximun tolerated dose (MTD) of FF-10850 | 4 years
  MTD is defined as the next lower dose of a cohort where patients experienced a DLT
Determine recommended Phase 2 dose (RP2D) FF-10850 | 4 years
  The highest dose level below the dose level eliciting DLT in ≥ 2 patients will be declared the MTD. The RP2D will be chosen based on the MTD or on PK and biological activity if an MTD has not been determined.

SECONDARY OUTCOMES:
Characterize the pharmacokinetics (PK) of FF-10850 in plasma: Cmax | 4 years
  Measurement of maximum plasma concentration
Characterize the pharmacokinetics (PK) of FF-10850 in plasma: tmax | 4 years
  Measurement of time to reach Cmax
Characterize the pharmacokinetics (PK) of FF-10850 in plasma: t1/2 | 4 years
  Measurement of the elimination half-life
Characterize the pharmacokinetics (PK) of FF-10850 in plasma: AUC | 4 years
  Measurement of the area under the curve of plasma concentration versus time profile
Characterize the pharmacokinetics (PK) of FF-10850 in plasma: MRT | 4 years
  Measurement of the mean residence time adjusted for duration of infusion
Characterize the pharmacokinetics (PK) of FF-10850 in plasma: CL | 4 years
  Measurement of the total plasma clearance
Characterize the pharmacokinetics (PK) of FF-10850 in plasma: Vss | 4 years
  Measurement of the steady-state volume of distribution for total topotecan
Determine objective response rate (ORR) | 4 years
  classified for solid tumors via RECIST v.1.1
Determine the duration of response (DOR) | 4 years
  Duration of Response is calculated from the date of first response to the date of progression or death.
Determine the time to progression (TTP) | 4 years
  Time to progression is calculated from the date of first treatment to the date of first progression
Evaluate progression-free survival (PFS) | 4 years
  Progression-free survival will be calculated from the date of first treatment to the date of progression or death
Evaluate overall survival (OS) (expansion cohorts only) | 4 years
  Overall survival will be calculated from the date of first treatment to the date of death from any cause; patients who do not experience death will be censored at the last follow-up time.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - HonorHealth, Scottsdale, Arizona
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Dana Farber Cancer Institute (DFCI), Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shimoyama S, Okada K, Kimura T, Morohashi Y, Nakayama S, Kemmochi S, Makita-Suzuki K, Matulonis UA, Mori M. FF-10850, a Novel Liposomal Topotecan Achieves Superior Antitumor Activity via Macrophage- and Ammonia-Mediated Payload Release in the Tumor Microenvironment. Mol Cancer Ther. 2023 Dec 1;22(12):1454-1464. doi: 10.1158/1535-7163.MCT-23-0099. PMID 37683276